CLINICAL TRIAL: NCT02860819
Title: Phase II Study of Gemcitabine, Carboplatin and VELIPARIB (ABT-888) in Refractory Testicular Germ Cell Cancer
Brief Title: Study of Gemcitabine, Carboplatin and VELIPARIB (ABT-888) in Refractory Testicular Germ Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCTSK004
Record Dates: First submitted 2016-07-14; First posted 2016-08-09 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2020-12

CONDITIONS: Testicular Cancer
Keywords: Multiple relapsed/refractory testicular germ cell tumors; PARP inhibition; Chemotherapy; Gemcitabine; Carboplatin
MeSH Terms: conditions — Testicular Neoplasms | interventions — veliparib; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine, Carboplatin, Veliparib (Experimental): Gemcitabine 800mg/m2 day 1 and 8 every 3 weeks; Carboplatin AUC = 4, day 1, every 3 weeks, Veliparib 250mg bid day continuously.
  Interventions: Drug: Veliparib; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Veliparib — Veliparib 250mg BID, continuously
  Other Names: ABT-888
Drug: Gemcitabine — Gemcitabine 800mg/m2, day 1 and 8
Drug: Carboplatin — Carboplatin AUC = 4, day 1

SUMMARY:
This is a proof-of-concept study to define efficacy of gemcitabine, carboplatin and VELIPARIB (ABT-888) in patients with refractory germ cell tumors (GCTs). PARP proteins are involved in base excision repair (BER), one of the major DNA repair system in cells and PARP is overexpressed in testicular GCTs (TGCTs) compared to normal testis and data suggest that PARP overexpression is early event in TGCTs development. Patients with low PARP expression in primary tumour had non-significantly better OS compared to patients with high PARP expression (5-year OS 89.2% vs 78.7%; HR=0.50, 95% CI 0.21 to 1.17, p=0.12). The aim of this study is to evaluate PARP inhibitor VELIPARIB in combination with gemcitabine, carboplatin in patients with refractory germ cell tumors (GCTs).

DETAILED DESCRIPTION:
PARP proteins are involved in base excision repair (BER), one of the major DNA repair system in cells. Recently, it was showed that PARP inhibitors have striking efficacy in patients with BRCA1 deficient or triple negative breast cancer in monotherapy or in combination with cisplatin based chemotherapy, without increased systemic toxicity. Pertubations affecting homologous recombination (HR) involved in DNA repair are associated with higher probability of response to PARP inhibitors. Inactivation of PTEN, tumor suppressor protein, is associated with defects in HR and response to PARP inhibitors.

Recently, PARP expression was evaluated in TGCTs. It was showed that PARP is overexpressed in testicular germ cell tumours compared to normal testis and PARP overexpression is early event in TGCTs development. Patients with low PARP expression in primary tumour had non-significantly better OS compared to patients with high PARP expression (5-year OS 89.2% vs 78.7%; HR=0.50, 95% CI 0.21 to 1.17, p=0.12).Loss of the tumor suppressor gene PTEN marks the transition from intratubular germ cell neoplasias (ITGCN) to invasive germ cell tumors. In the testis, PTEN was abundantly expressed in germ cells whereas it was virtually absent from 56% of seminomas as well as from 86% of embryonal carcinomas and virtually all teratomas. On the contrary, ITGCN intensely expressed PTEN, indicating that loss of PTEN expression is not in early event in testicular tumor development, but is associated with progression of disease. Previously, it was showed, that testicular germ cell tumors cell lines have low activity of proteins involved in nuclear excision repair (NER) and it is assumed that low NER activity is related to the favorable response of testis tumors to cisplatin-based chemotherapy.

Gemcitabine and carboplatin showed activity in refractory TGCTs. Recently, maximal tolerated dose of Veliparib (ABT-888) with gemcitabine and carboplatin was established.

Based on aforementioned data, there is strong rationale to inhibit PARP in TGCT. Inactivation of PARP by Veliparib along with defects of homologous recombination due to PTEN inactivation in GCTs and low activity of nucleotide excision repair system will dramatically increase antitumor effect gemcitabine and carboplatin in patients with progressing or relapsing germ cell cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Men aged 18 years or older
3. ECOG performance status: 0-1,
4. Histologically confirmed extracranial primary germ cell cancer, seminoma, or nonseminoma
5. Rising serum markers (i.e., alpha-fetoprotein and human chorionic gonadotropin) on sequential measurement or biopsy-proven unresectable germ cell cancer
6. Refractory GCTs e.g. patients relapsing after high-dose chemotherapy or for patients non fit enough for high-dose chemotherapy
7. Primary mediastinal GCTs in first relapse
8. Patient's disease must not be amenable to cure with either surgery or chemotherapy in the opinion of investigator,
9. Measurable disease radiologically
10. Adequate hematologic function defined by ANC > 1500/mm3, platelet count > 100 000/mm3 and hemoglobin level > 9g/dl.
11. Adequate liver function defined by a total bilirubin level < 1.5 ULN, and ALT, AST < 3 ULN or < 5 in case of liver metastases. For subjects with Gilbert's syndrome bilirubin > 1.5 × ULN is allowed if no symptoms of compromised liver function are present
12. Adequate renal function: measured or calculated (by Cockcroft formula) creatinine clearance > 50 ml/min. Cockcroft formula: CLcr = [(140-age) x weight(Kg)]/[72 x creatinine (mg/dl)]
13. At least 4 weeks must have elapsed since the last radiotherapy and/or chemotherapy before study entry,
14. At least 4 weeks must have elapsed since the last major surgery
15. Complete recovery from prior surgery, and/or reduction of all adverse events from previous systemic therapy or radiotherapy to grade 1,
16. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Exclusion Criteria:

1. Patients who do not fit inclusion criteria
2. Other prior malignancy except successfully treated nonmelanoma skin cancer
3. Prior PARP1 inhibitor
4. Other concurrent approved or investigational anticancer treatment, including surgery, radiotherapy, chemotherapy, biologic-response modifiers, hormone therapy, or immunotherapy
5. Female patients
6. Patients infected by the Human Immunodeficiency Virus (HIV)
7. Patients with other severe acute or chronic medical condition, or laboratory abnormality that would impair, in the judgment of investigator, excess risk associated with study treatment, or which, in judgment of the investigator, would make the patient inappropriate for entry into this study
8. Inability of oral intake, or drug absorption (e.g. malabsorption syndrome)
9. Hypersensitivity to any compound of the drug
10. Sexually active men not using highly effective birth control if their partners are women of child-bearing potential
11. Patients with history of or current CNS metastasis
12. Patients with history of seizures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that will be free of disease progression according to RECIST criteria 12-months after the first administration of the treatment. | 12-months
  Percentage of patients that will be free of disease progression according to RECIST criteria 12-months after the first administration of the treatment.

SECONDARY OUTCOMES:
Response rate | 6-weeks
  Response rate as measured by RECIST 1.1
Median overall survival | 12 months
  Median overall survival. Overall survival will be measured from the date of first administration of the treatment until death or date of last follow-up.
Median progression-free survival | 12-months
  Median progression-free survival. Progression-free survival will be measured from the date of first administration of the treatment until progression, death or date of last follow-up.
Frequency of grade III and IV adverse events | 3-weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, Assoc.Prof, Study Chair — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mego M, Svetlovska D, Reckova M, Angelis D, Kalavska K, Obertova J, Palacka P, Rejlekova K, Sycova-Mila Z, Chovanec M, Mardiak J. Gemcitabine, carboplatin and veliparib in multiple relapsed/refractory germ cell tumours: The GCT-SK-004 phase II trial. Invest New Drugs. 2021 Dec;39(6):1664-1670. doi: 10.1007/s10637-021-01130-5. Epub 2021 May 29. PMID 34052929